CLINICAL TRIAL: NCT07019441
Title: A Daily-Activity-Focused, Strategy-Based Educational Programme for Informal Dementia Carers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIU Karen, Prof., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HongKongPU_Dementia carer edu
Record Dates: First submitted 2025-05-25; First posted 2025-06-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Informal Caregivers
Keywords: informal carers; dementia; carer education; daily activities
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blind assessors will collect data and they do not have any knowledge about participants' group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily-Activity-Focused, Strategy-Based Educational Program (Experimental): The intervention / experimental group will have one face-to-face education session, three follow-up telephone support sessions and a final home visit or phone call. Strategies to assist people with dementia with daily activities are compiled into the Carer Strategies Package. Healthcare professionals will deliver the program and work collaboratively with the informal carers to identify issues that arise during caregiving and problem-solve using the strategies included in the package.
  Interventions: Other: Daily-Activity-Focused, Strategy-Based Educational Program
- Usual Support Program (Active Comparator): The control group will receive emotional support from healthcare professionals on the caring issues raised. They will be provided with resource information about dementia and care. It will also include the same number of sessions as the experimental group in which carers will discuss the caring difficulties and possible solutions with the healthcare professionals as well as access to online resources.
  Interventions: Other: Usual Carer support

INTERVENTIONS:
Other: Daily-Activity-Focused, Strategy-Based Educational Program — The proposed Educational Program will have one face-to-face education session and three follow-up telephone support sessions. Strategies to assist the people with dementia with daily activities, developed from our prior work, have been compiled into a Strategies Package. Healthcare professionals will deliver the program and work collaboratively with the carers to identify issues that arise during caregiving and problem-solve using the strategies included in the package. Carers are provided with support and are encouraged to locate an appropriate strategy using the Strategies Package to help them assist in a daily task in which they want their care recipient to engage.
  Arms: Daily-Activity-Focused, Strategy-Based Educational Program
Other: Usual Carer support — This group will receive emotional support from trainers on the caring issues raised. It will include the same number of sessions as in the experimental group.
  Arms: Usual Support Program

SUMMARY:
This study will assess the impact of the Dementia Carer Education Programme on the caregiving burden of informal dementia carers.

Ninety informal dementia carers along with their care-recipients will be recruited and randomised to the experimental and control groups. All recruited dementia carers in the experimental group will receive the Dementia Carer Education Programme and the control group will receive usual carer support, both including one face-to-face education session and four follow-up sessions over 7 weeks. Caregiving burden will be assessed after receiving the programme. Statistical analysis of caregiving burden will follow the intention-to-treat principle, employing paired t-tests and linear modelling.

DETAILED DESCRIPTION:
Objective. To investigate the effectiveness of a Daily-Activity-Focused, Strategy-Based Educational Program for informal carers when helping people with dementia with daily activities using a randomised controlled trial design.

Participants. This part will recruit 'trainers' to deliver the program. Six healthcare professionals will recruit a total of 15 carers. A total of 90 carers will then be recruited.

Block randomisation will be used to randomise carers of each participating healthcare professional such that an equal number of carers are assigned to the 'Daily-Activity-Focused, Strategy-Based Educational Program' experimental or the 'usual carer support' control groups. Training will be provided to all participating healthcare professionals to deliver either the experimental or control program to carers.

All six healthcare professionals will have over five years of experience working with people with dementia and their carers.

Dyads (care-recipients and their carers) will be recruited. The inclusion criteria will be as follows: (1) the care-recipient has dementia; (2) the carer is the primary carer and assumes responsibility for the care-recipient; (3) the carer is at least 18 years old; and (4) primary care takes place at home. The exclusion criteria will be as follows: (1) the care-recipient's impairments in daily activities are primarily due to medical conditions other than dementia, such as stroke, and (2) the carer has a cognitive impairment that may hinder their understanding of and engagement with the programs.

Using the change in carer burden as the outcome, 45 dyads in each group, which would allow for a 10% estimated dropout, will give a power of 80%, an effect size of 0.25, and an alpha value of 0.05.

Daily-Activity-Focused, Strategy-Based Educational Program. Our pilot studies indicate that the proposed Educational Program will have one face-to-face education session and three follow-up telephone support sessions. Strategies to assist people with dementia with daily activities, developed from our prior work, have been compiled into a Strategies Package. Healthcare professionals will deliver the program and work collaboratively with the carers to identify issues that arise during caregiving and problem-solve using the strategies included in the package. Carers are provided with support and are encouraged to locate an appropriate strategy using the Strategies Package to help them assist in a daily task in which they want their care recipient to engage.

Usual Carer support. This group will receive emotional support from trainers on the caring issues raised. It will include the same number of sessions as in the experimental group.

Data collection. The demographic information of the participating healthcare professionals, care-recipients and carers will be collected before the program. Medical and functional data on the care-recipients will be collected. The outcome measures used will be administered to the carers before and immediately after the program.

Outcome measures. The primary outcome measures include (1) Zarit Burden Inventory (ZBI). The secondary outcome measures include (2) Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale (ADCS-ADL); and (3) Adult Carer Quality of Life Questionnaire (AC-QoL). Other secondary outcome measures include the number of Emergency Department visits, hospital admissions and length of stay, aged care facility admissions and length of stay. They will be recorded six months after the program.

Statistical analysis. Descriptive statistics will be reported for all data collected. Two-way repeated-measure analysis of variance (ANOVA) will be used to compare the primary outcomes collected pre- and post-program between the two groups. The difference in the secondary outcomes between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. the care-recipient has dementia;
2. the carer is the primary carer and assumes responsibility for the care-recipient;
3. the carer is at least 18 years old; and
4. primary care takes place at home.

Exclusion Criteria:

1. the care-recipient's impairments in daily activities are primarily due to medical conditions other than dementia, such as stroke, and
2. the carer has a cognitive impairment that may hinder their understanding of and engagement with the programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Zarit Burden Inventory | From enrollment to the end of program at 7 weeks
  Zarit Burden Interview (ZBI) is a 22-question, paper-based self-reported questionnaire developed to be used with carers of people with dementia within the community. The overall score interpretation ranges from zero to 88, from 'little or no burden' to 'severe burden'.

SECONDARY OUTCOMES:
Adult Carer Quality of Life Questionnaire | From enrollment to the end of program at 7 weeks
  Adult Carer Quality of Life Questionnaire (AC-QoL) is a 40-question, paper-based self-reported instrument used to screen for quality of life. The tool uses sub-scales including support for caring, caring choice, caring stress, money matters, personal growth, sense of value, ability to care and carer satisfaction, highlighting the holistic impact of caring on an individual. The sub-scales are similarly scored from 'low reported quality of life' to 'high reported quality of life', with scores ranging from zero to 120.
Alzheimer's Disease Cooperative Study- Activities of Daily Living Scale | From enrollment to the end of program at 7 weeks
  The Alzheimer's Disease Cooperative Study- Activities of Daily Living Scale is a 23-item paper-based questionnaire reported by the carer about the care-recipient's performance covering a range of daily activities. The scoring ranges from zero to 78, from profound severity to typical performance.

OTHER OUTCOMES:
Number of Emergency Department visits | Six months after the educational program
  They reflect the potential effect of the educational program on the hospital admission of persons with dementia.
Number of hospital admissions | Six months after the educational program
  They reflect the potential effect of the educational program on the hospital admission of persons with dementia.
length of hospital stay | Six months after the educational program
  They reflect the potential effect of the educational program on the length of hospital stay of persons with dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Karen P. Y. Liu, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The project is currently collecting pilot data only, and the results will be used to apply for external funding.

REFERENCES:
- [Background] Burridge G, Amato C, Bye R, Basic D, Ni Chroinin D, Hill S, Howe K, Liu KPY. Strategies adopted by informal carers to enhance participation in daily activities for persons with dementia. Australas J Ageing. 2024 Dec;43(4):683-691. doi: 10.1111/ajag.13341. Epub 2024 May 28. PMID 38804160
- [Background] Amato C, Burridge G, Basic D, Huynh D, Gibbons E, Ni Chroinin D, Liu KPY. Assistance provided in daily tasks and difficulty experienced by caregivers for people living with dementia. Aust Occup Ther J. 2021 Jun;68(3):236-245. doi: 10.1111/1440-1630.12720. Epub 2021 Feb 2. PMID 33533025